CLINICAL TRIAL: NCT06729320
Title: A Randomized Controlled, Open, Single-center Clinical Study Evaluating the Efficacy and Safety of Umbilical Cord Blood Mononuclear Cells in Patients with Refractory Immune Effector Cell-related Hemocytopenia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing GoBroad Hospital (Other)
Responsible Party: Principal Investigator, Kai Hu, Principal Investigator, Beijing GoBroad Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCB-MNCs-2024
Record Dates: First submitted 2024-12-08; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Refractory Immune Effector Cell-related Hemocytopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional hematopoietic recovery therapy (Active Comparator): Conventional hematopoietic recovery therapy including but not limited to G-CSF, TPO, TPO receptor agonists, transfusions of red blood cells, platelets, etc.
  Interventions: Combination Product: Conventional hematopoietic recovery therapy
- Conventional hematopoietic recovery therapy+Umbilical cord blood mononuclear cells (Experimental): Umbilical cord blood mononuclear cells are obtained from umbilical cord blood by density gradient centrifugation
  Interventions: Biological: Umbilical cord blood mononuclear cells; Combination Product: Conventional hematopoietic recovery therapy

INTERVENTIONS:
Biological: Umbilical cord blood mononuclear cells — Intravenous infusion of UCB-MNCs (3×10^8/ time, once a week, four times in total)
  Arms: Conventional hematopoietic recovery therapy+Umbilical cord blood mononuclear cells
Combination Product: Conventional hematopoietic recovery therapy — Including but not limited to G-CSF, TPO, TPO receptor agonists, transfusions of red blood cells, platelets, etc.

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of umbilical cord blood mononuclear cell in the treatment of refractory immune effector cell-related hemocytopenia by observing the efficacy related factors and adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old (including boundary values), gender is not limited
2. ECOG score 0-2 points
3. Expected survival ≥6 months
4. Patients who have received immune effector cell therapy (marketed CAR-T cell therapy or dual antibody therapy) (no target), have grade 3-4 hemocytopenia after treatment, and do not recover to grade 2 within 3 weeks after conventional treatment. Defined as follows:

1) The neutrophils again decreased to grade ≥3 within 1 week after G-CSF discontinuation, or 2) Unable to detach from red blood cell or platelet transfusion (infusion time less than one week requires re-infusion) (5) Understand the research protocol and sign the informed consent voluntarily

Exclusion Criteria:

1. Patients who intend to undergo autologous hematopoietic stem cell transfusion or have undergone autologous hematopoietic stem cell transfusion
2. Significant lack of compliance to complete the study plan (such as suffering from uncontrolled mental illness, etc.)
3. Allergy or known allergy to any drug active ingredients, excipients, and blood products or preparations included in this study
4. Pregnancy, breastfeeding, planning pregnancy, or unwillingness to use effective contraception as required by research
5. There are other conditions that researchers believe are not suitable for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The recovery time of neutrophils | 1 year
  On the first day after discontinuing G-CSF, the neutrophil count remained above 1.0 × 10^9/L for 7 consecutive days
The recovery time of platelet | 1 year
  Starting from the second day of the most recent platelet transfusion, the first day of platelet count>50 × 10^9/L lasting for 7 days
Safety of infusion | 1 year
  Acute allergies or infections related to umbilical cord blood mononuclear cell infusion, as well as shock and other infusion related reactions symptoms including but not limited to chills, fever, CRP, PCT, etc

SECONDARY OUTCOMES:
Recovery of hemoglobin levels after infusion | 1 year
  Hemoglobin content in blood routine examination
Immune function reconstruction indicators at 1, 3, 6, and 12 months after transfusion | 1, 3, 6, and 12 months
  Including but not limited to CD3, CD4, CD8, CD19, etc. in lymphoid subgroups
Overall survival rate | 2 and 5 year
  The proportion of participants who survived during the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing GoBroad Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No